CLINICAL TRIAL: NCT01093807
Title: Randomized, Parallel Group, Double-blind Trial to Evaluate Different Dose Combinations of Lercanidipine and Enalapril in Comparison With Each Component Administered Alone and With Placebo in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of Lercanidipine and Enalapril in Patients With Essential Hypertension
Acronym: FELT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Barbara Bettini - Clinical Project Leader, Medical Department
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: REC 15/2375-IT-CL 0336
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Essential Hypertension
Keywords: Hypertension; Lercanidipine; Calcium antagonist; Enalapril
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — lercanidipine; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Lercanidipine 10 mg (Experimental)
  Interventions: Drug: Lercanidipine
- Lercanidipine 20 mg (Experimental)
  Interventions: Drug: Lercanidipine
- Enalapril 10 mg (Experimental)
  Interventions: Drug: Enalapril
- Enalapril 20 mg (Experimental)
  Interventions: Drug: Enalapril
- Lercanidipine 10 mg/Enalapril 10 mg (Experimental)
  Interventions: Drug: Lercanidipine + Enalapril
- Lercanidipine 10mg/Enalapril 20 mg (Experimental)
  Interventions: Drug: Lercanidipine + Enalapril
- Lercanidipine 20mg/Enalapril 10 mg (Experimental)
  Interventions: Drug: Lercanidipine + Enalapril
- Lercanidipine 20mg/Enalapril20mg (Experimental)
  Interventions: Drug: Lercanidipine + Enalapril

INTERVENTIONS:
Drug: Placebo — once daily for 10 weeks
  Arms: Placebo
Drug: Lercanidipine — 10 mg once daily for 10 weeks
  Arms: Lercanidipine 10 mg
Drug: Lercanidipine — 20 mg once daily for 10 weeks
  Arms: Lercanidipine 20 mg
Drug: Enalapril — 10 mg once daily for 10 weeks
  Arms: Enalapril 10 mg
Drug: Enalapril — 20 mg once daily for 10 weeks
  Arms: Enalapril 20 mg
Drug: Lercanidipine + Enalapril — 10/10 mg once daily for 10 weeks
  Arms: Lercanidipine 10 mg/Enalapril 10 mg
Drug: Lercanidipine + Enalapril — 10/20 mg once daily for 10 weeks
  Arms: Lercanidipine 10mg/Enalapril 20 mg
Drug: Lercanidipine + Enalapril — 20/10 mg once daily for 10 weeks
  Arms: Lercanidipine 20mg/Enalapril 10 mg
Drug: Lercanidipine + Enalapril — 20/20 mg once daily for 10 weeks
  Arms: Lercanidipine 20mg/Enalapril20mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of various dosage combinations of lercanidipine (10 and 20 mg)and enalapril (10 and 20 mg) in comparison with their respective components and with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Office Blood Pressure (BP): Sitting diastolic blood pressure (SDBP)100-109 mmHg (inclusive) and sitting systolic blood pressure (SSBP) < 180 mmHg after a 2 week placebo run-in period
* Home Blood Pressure: diastolic blood pressure (DBP)at home ≥ 85 mmHg in the last week of the placebo run-in period
* Normal Electrocardiogram (ECG), first degree Atrioventricular block or other changes not considered clinically significant

Exclusion Criteria:

* Secondary or severe hypertension
* History of cerebro- or cardiovascular complications
* Type 1 or Type 2 diabetes on drug treatment
* Severe renal or hepatic insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1039 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sitting diastolic blood pressure (SDBP) | after 10 weeks

SECONDARY OUTCOMES:
Change from baseline in sitting systolic blood pressure (SSBP) | after 10 weeks
Safety parameters: adverse events, heart rate, laboratory tests physical examination | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Mancia, Prof, Study Chair — Clinica Medica Ospedale S. Gerardo Università Milano Bicocca Italy
Locations (1):
- Hôpital de la Pitié-Salpétrière, Paris, France

REFERENCES:
- [Derived] Mancia G, Omboni S, Chazova I, Coca A, Girerd X, Haller H, Parati G, Pauletto P, Pupek-Musialik D, Svyshchenko Y; FELT Study Group. Effects of the lercanidipine-enalapril combination vs. the corresponding monotherapies on home blood pressure in hypertension: evidence from a large database. J Hypertens. 2016 Jan;34(1):139-48. doi: 10.1097/HJH.0000000000000767. PMID 26630216